CLINICAL TRIAL: NCT04596969
Title: The Effect of Soluble Fiber Dextrin on Subjective and Physiological Markers of Appetite: a Randomized Trial
Brief Title: The Effect of Soluble Fiber Dextrin on Subjective and Physiological Markers of Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SFDISU
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Appetitive Behavior
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Intervention Model Description: Human subjects
Who Masked: Participant, Investigator
Masking Description: Material was provided in coded plain packaging. Participants and researchers were unaware of what was being received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- SFD Tapioca 20g (Experimental): 20g soluble fiber dextrin derived from tapioca
  Interventions: Other: Soluble Fiber Dextrin
- SFD Tapioca 40g (Experimental): 40g soluble fiber dextrin derived from tapioca
  Interventions: Other: Soluble Fiber Dextrin
- SFD corn 20g (Experimental): 40g soluble fiber dextrin derived from corn
  Interventions: Other: Soluble Fiber Dextrin
- SFD corn 40g (Experimental)
  Interventions: Other: Soluble Fiber Dextrin
- Control (Placebo Comparator): Maltodextrin
  Interventions: Other: Soluble Fiber Dextrin

INTERVENTIONS:
Other: Soluble Fiber Dextrin — Ingredient based on resistant starch

SUMMARY:
This study examines the effect of soluble fiber dextrin on food intake, appetite, and physiological markers of appetite. Adults aged 18-45 years with a BMI were recruited for this study. Participants were given two doses of SFD in the morning and appetite, food intake and physiological markers of appetite were measured over 10 years.

DETAILED DESCRIPTION:
Overweight and obesity are leading health problems. The study investigates the effect of a food ingredient from two different sources at two different doses on food intake and appetite markers over a 10 hour period. All participants reported to the laboratory first thing in the morning and remained in the laboratory until after their evening meal. A fixed breakfast was served but the participants were free to eat as much as they liked at lunch and dinner. Blood was taken at regular intervals during the day and assayed for glucose and several hormones related to appetite. Subjective measures of appetite were also collected over the 10 hour test session.

ELIGIBILITY:
Inclusion Criteria:

BMI 19.9 - 29.9 Aged 18-45 Find the study foods to be palatable

Exclusion Criteria:

Weight change > 3kg in the past three months Do not regularly consume snacks Presence or history of GI disorders Restrained eater Used medication that influences appetite

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Food intake | 10 hours
  Food intake measured at lunch and evening meal.

SECONDARY OUTCOMES:
Appetite | 10 hours
  Subjective appetite measures using questionnaires at regular intervals over 10 hours,
CCK | 10 hours
  Plasma CCK measured at regular intervals over 10 hours.
GLP-1 | 10 hours
  Plasma GLP-1 measured at regular intervals over 10 hours.
PYY3-36 | 10 hours
  Plasma PYY3-36 measured at regular intervals over 10 hours.
Breath Hydrogen | 10 hours
  Breath hydrogen measured at regular intervals over 10 hours.

IPD SHARING:
Plan to Share IPD: No